CLINICAL TRIAL: NCT04134026
Title: Phase 4, Multicenter, Randomized, Open-Lable, Active-Controlled Study of the Efficacy and Safty of HIF-PHI for the Treatment of Anemia and Risks of Cardiovascular and Cerebrovascular Events in Incident-Dialysis Patients
Brief Title: Evaluate the Efficacy and Safety of HIF-PHI for the Treatment of Anemia and Risks of Cardiovascular and Cerebrovascular Events in ESRD Newly Initiated Dialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Hong Liu, Director of Department of Nephrology, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSU-SXH-CT-2019-015
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Anemia in Incident Dialysis Patients
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIF-PHI (Experimental): HIF-PHI will be dosed orally three times a week.
  Interventions: Drug: HIF-PHI
- Epoetin alfa (Active Comparator): Epoetin alfa wull be disoensed per the package insert or the country-specific product labeling.
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: HIF-PHI — Drug will be dosed orally three times a week.
  Arms: HIF-PHI
Drug: Epoetin Alfa — The drug will be dispensed per the package insert or the country-specific product labeling.
  Other Names: Epogen
  Arms: Epoetin alfa

SUMMARY:
The purpose of the study is to determin whether HIF-PHI is safe and effective in the treatment of anemia and meanwhile reduces the risk of cardiovascular and cerebrovascular events in patients who have just initiated dialysis.

DETAILED DESCRIPTION:
There is a screening period of up to 2 weeks, a treatment period of a minimum of 52 weeks and a maximum of approximately up to 3 years after last patient is randomized. A total of up to 400 patients will be randomized in a 1:1 ratio to receive either open-lable HIF-PHI or Active Control (Epoetin alfa).

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her legal guardian signs the informed consent
2. Age ≥18 years
3. Weight: 45-100 kg (included)
4. Patients with CKD end-stage renal disease received hemodialysis treatment ≤ 4 weeks, dialysis frequency was stable, kt / V ≥ 1.2, and planned to continue dialysis treatment during the study period
5. No iron deficiency.
6. No folate or Vitamin B12 deficiency.
7. No abnormal liver tests.
8. During the screening period, value of Hb is less than 10. 0 g / dl.

Exclusion Criteria:

1. Evidence of any clinically significant infection or active potential infection;
2. Active hepatitis or any of the following abnormalities (ALT ≥ 2 times the upper limit of normal value, AST ≥ 2 times the upper limit of normal value, DBIL ≥ 2 times the upper limit of normal value);
3. Patients with severe cardiovascular disease have had myocardial infarction, coronary artery bypass or PCI operation within 3 months prior to participating in the study.
4. Patients have experienced severe cerebrovascular diseases within 3 months prior to participating in the study: stroke; obvious neurological dysfunction after stroke;
5. Patients with active gastrointestinal bleeding occurred within 3 months prior to participating in the study.
6. Poor control of hypertension determined by the researchers;
7. Previous or current malignancies (except for excised non melanoma skin cancer and carcinoma in situ);
8. It is known to have blood system diseases (including congenital and postnatal diseases, such as thalassemia, Fanconi anemia, aplastic anemia, myelodysplastic syndrome, hemolytic anemia, coagulation dysfunction, etc.) or other causes of anemia (such as fecal occult blood positive gastrointestinal hemorrhage or hookworm disease, etc.) ;
9. Known autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, anti neutrophil cytoplasmic antibody associated vasculitis, etc.);
10. Any previous functional organ transplant or scheduled organ transplant or no kidney.
11. Elective surgery that is expected to result in significant blood loss during the study period.
12. Serum albumin < 25 g / L;
13. Within 8 weeks before administration on the first day, the patients were treated with androgen, deferoxamine, deferrone or deferestrol.
14. Life expectancy < 12 months;
15. Transfusion within 4 weeks before administration on day 1, or is expected.
16. Intravenous iron supplementation and / or unwillingness to stop intravenous iron injection during the screening period;
17. Patients with drug abuse or addiction;
18. Have received any test drug within 4 weeks before inclusion or plan to receive other drug tests during the trial;
19. Women who can become pregnant must use contraception. Men with sexual partners who can become pregnant must use birth control, unless the man agrees to use contraception.
20. Any medical condition, that in the opinion of the study doctor, may pose a safety risk to the patient, may confound efficacy or safety assessment, or may interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-10-19 (Estimated); Study Completion 2024-10-19 (Estimated)

PRIMARY OUTCOMES:
Mean Hemoglobin (Hb) change from baseline to average levels from Week 28 to Week 52. | Minimum of 52 weeks and maximum of up to 3 years after last subject is randomized
  For participants who did not have an available Hb value during the week 28-52 period, imputation rules were applied.
Proportion of subjects who achieve a Hb response during the first 24 weeks of treatment. | Week 0 to Week 24
  A Hb response is defined as:
  Hb ≥11.0g/dL and a Hb increase from baseline by ≥1.0g/dL in subjects whose baseline Hb >8.0g/dL, or Increase in Hb ≥2.0g/dL in subjects whose baseline Hb ≤8.0g/dL.
The incidence of cardiovascular and cerebrovascular events within 52 weeks. | Week 0 to Week 52
  Non fatal myocardial infarction, unstable angina, coronary artery bypass, coronary or peripheral vascular intervention, hospitalization due to heart failure, transient ischemic attack, stroke and death.

SECONDARY OUTCOMES:
All cause mortality | Minimum of 52 weeks and maximum of up to 3 years after last subject is randomized
  The incidence of death events.
BP effect 1: the proportion of subjects with increased hypertension | Week 0 to Week 27
  Blood pressure (BP) increased compared to pre-dialysis BP: the delta systolic BP ≥ 20 mmHg and systolic blood pressure ≥ 170 mmHg, or the delta diastolic BP ≥ 15 mmHg and diastolic BP ≥ 100 mmHg.
BP effect 2 | Week 28 to Week 52
  Mean BP change from baseline to average levels from Week 28 to Week 52.
The change of left ventricular structure | Weeks 12, 36, 52
  Standardized ECHO evaluates left ventricular volume index (ml/m2).
The change of left ventricular systolic function | Weeks 12, 36, 52
  Standardized ECHO evaluates left ventricular ejection fraction (%).
The change of right ventricular systolic function | Weeks 12, 36, 52
  Systolic lateral tricuspid annulus velocity (S') was measured by tissue Doppler.
The change of diastolic function | Weeks 12, 36, 52
  Left ventricular diastolic function was measured based on the integration of the ratio of early (E wave) and late (A wave) mitral inflow, mitral E wave deceleration time, E/e' ratio (e' being the tissue Doppler velocity of the medial annulus), E/A changes with Valsalva maneuver, and pattern of pulmonary vein flow. The data will be combine to report diastolic function.
Serum lipid parameters | Week 25 to Week 27
  Mean change in low-density lipoprotein (LDL) cholesterol.
Inflammatory evaluation 1 | Week 25 to Week 27
  Mean change level of CRP.
Inflammatory evaluation 2 | Week 25 to Week 27
  Mean change level of IL-2
Inflammatory evaluation 3 | Week 25 to Week 27
  Mean change level of IL-6
Inflammatory evaluation 4 | Week 25 to Week 27
  Mean change level of IL-17A

OTHER OUTCOMES:
Serum iron level | Week 0 to Week 27
  Mean change of iron from baseline to level at the 27th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278